CLINICAL TRIAL: NCT04533633
Title: German Multicentre Registry to Evaluate the Technical Feasibilty of Epicardial Collateral Connections in CTO PCI
Brief Title: German Epicardial Collateral CTO Registry
Acronym: EPIC
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitätsmedizin Mannheim (Other)
Collaborators: University Heart Center Freiburg - Bad Krozingen (Other)
Responsible Party: Principal Investigator, Michael Behnes, Principal Investigator, Universitätsmedizin Mannheim
Other Study IDs: 2017-838R-MA
Record Dates: First submitted 2020-08-23; First posted 2020-08-31 (Actual); Last update posted 2020-09-01 (Actual); Status verified 2020-08

CONDITIONS: Coronary Artery Disease; Chronic Total Occlusion; Percutaneous Coronary Intervention
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Retrograde Percutaneous Coronary Intervention of Chronic Total Occlusion — Retrograde CTO-PCI using epicardial collateral connections

SUMMARY:
The EPIC registry is an observational multicentre registry evaluating the technical feasibility of retrograde CTO-PCI using epicardial collateral connections. It will evaluate the frequency, effectiveness, safety and outcomes of patients who underwent CTO-PCI using this approach. The EPIC registry retrieves data from CTO centres across Germany.

DETAILED DESCRIPTION:
The EPIC registry is the first German-wide observational multicentre registry evaluating the technical feasibility, clinical success and safety of retrograde CTO-PCI using epicardial collateral connections. The EPIC registry retrieves data from CTO centres across Germany. All patients will be followed-up to 30 days after inclusion.

ELIGIBILITY:
Inclusion Criteria:

* All patients undergoing retrograde CTO-PCI using epicardial collateral connections during daily clinical practice.

Exclusion Criteria:

* None.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: EPIC will observationally evaluate all patients undergoing retrograde CTO-PCI using epicardial collateral connections during daily clinical practice from German CTO centres.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of technically successful retrograde CTO-PCI using epicaridal collaterals | 30 days
  defined as the rate of successful CTO-PCI with reestablished antegrade coronary flow (thrombolysis in myocardial infarction (TIMI) flow III) with less than residual stenosis of 50%.

SECONDARY OUTCOMES:
Rate of clinically successful retrograde CTO-PCI using epicaridal collaterals | 30 days
  Clinical success is defined as the rate of successful CTO-PCI by technical success without MACCE and without major periprocedural complications, including pericardial tamponade and contrast induced dialysis.
Rate of failed retrograde CTO-PCI using epicaridal collaterals | 30 days
  is defined as the rate of CTO-PCI without technical success defined as residual stenosis >50% (by visual estimation) and TIMI flow grade <3 after CTO-PCI.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Mannheim, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided